CLINICAL TRIAL: NCT03481374
Title: Cardiovascular Autonomic Neuropathy in Patients With Type 1 Diabetes Mellitus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, prof. dr., Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CVDIABMEL-1
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subjects with Type 1 Diabetes mellitus (Active Comparator): Type 1 diabetes patients without cardiovascular disease undergo autonomic function testing
  Interventions: Diagnostic Test: autonomic function testing
- Healthy controls (Placebo Comparator): healthy people without known disease undergo autonomic function testing
  Interventions: Diagnostic Test: autonomic function testing

INTERVENTIONS:
Diagnostic Test: autonomic function testing — autonomic function testing, ergospirometry, three questionnaires
  Other Names:
  * The autonomic function tests consist of five tests:
    * The Valsalva maneuver
    * The isometric handgrip test
    * The deep breathing test
    * The cold pressor test
    * A short head-up tilt test
  * A maximal ergospirometry
  * Three questionnaires:
    * EQ-5D-3L: quality of life
    * IPAQ: capacity to do physical activities

SUMMARY:
testing of autonomic function and relationship with exercise and Qol in diabetic patients and controls

DETAILED DESCRIPTION:
Cardiovascular autonomic neuropathy is a common (sub)clinical symptom in persons with type 1 diabetes mellitus. Subjects in this non-commercial, monocentric, interventional study undergo autonomic function tests, a maximal ergospirometry and three questionnaires about the quality of life (EQ-5D-3L), the capacity to do physical activities (IPAQ) and the experience of possible symptoms of autonomic dysfunction in daily life (SCOPA-AUT). In this way the influence of type 1 diabetes mellitus on the quality of life, the exercise capacity and the autonomic function can be studied.

The primary aim of this study investigates the potential correlations between the severity of diabetic cardiovascular autonomic neuropathy (DCAN) and both the quality of life and the exercise capacity. As a secondary aim, the influences of gender, age, number of years since diagnosis of type 1 diabetes mellitus, VO2 max predicted, maximal heart rate during exercise, minimal heart rate in rest, maximal RER (Respiratory exchange ratio) and relevant interaction terms are studied.

In total 52 test subjects with type 1 diabetes mellitus and 27 matched control subjects are selected to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (only for the group of subjects with diabetes mellitus)
* At least two years with diagnosis of type 1 diabetes mellitus
* Subject is in a stable condition
* No hospitalization for any reason in the past three months
* 18 years or older
* Being capable of doing physical activities
* Understand the study design and the informed consent
* Sign the informed consent
* No simultaneously participation to another study
* Being capable of moving to the study center

Exclusion Criteria:

* Uncontrolled hypertension, atrial fibrillation and other cardiovascular conditions
* Severe lung disease
* Muscle deficiency
* Medication with influence on the autonomic nervous system:

  * Beta blockers
  * Alfa blockers
  * Antidepressants
  * Non-catecholamines
  * (anti) cholinergic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
VO2 max | day 1
  peak oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: Renee De Busser, student, Study Chair — Hasselt University; Anika Nys, student, Study Chair — Hasselt University; Paul Dendale, prof. dr., Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided